CLINICAL TRIAL: NCT01510574
Title: A Study of Self-administered Misoprostol to Prevent Bleeding After Childbirth in the Community (MamaMiso)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: University of Liverpool (Other); Liverpool School of Tropical Medicine (Other); Makerere University (Other); Mbale Regional Referral Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3002
Record Dates: First submitted 2012-01-04; First posted 2012-01-16 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage, PPH, misoprostol
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- misoprostol (Active Comparator): 3 tablets of 200mcg misoprostol self-administered following home birth, taken orally immediately after delivery of baby
  Interventions: Drug: Misoprostol
- placebo (Placebo Comparator): 3 tablets of placebo resembling misoprostol self-administered following home birth, taken orally immediately after delivery of baby
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Misoprostol — 3 x 200mcg tablets of oral misoprostol
  Arms: misoprostol
Drug: placebo — 3 x placebo tablets resembling misoprostol taken orally
  Arms: placebo

SUMMARY:
Postpartum hemorrhage (PPH) is a major cause of maternal death in the developing world. An important strategy in the prevention of deaths is the use of uterotonic drugs for PPH prophylaxis. Misoprostol has been recognized as an option for preventing PPH as it is economical, heat stable, has a long shelf-life, and can be taken orally.

The investigators envisage that the use of self administered misoprostol after home births among mothers would be associated with a peri-partum fall in hemoglobin value of over 20% (the outcome of a fall of 2g/dl will also be tested in the pilot).

The objective of the main study will be to assess the effectiveness and safety of antenatal administration of misoprostol tablets (600mcg) for self administration immediately following home delivery for the prevention of postpartum haemorrhage. The objectives of the pilot study are to test the integrity of the study protocol, to test the randomization procedure, to assess the acceptability of the intervention, to test the logistics of follow-up, to test the data collection forms, to validate the quality of life questionnaire in this population and to determine the recruitment rate to help study planning.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women living in the recruitment villages of Mbale district at >34 weeks gestation

Exclusion Criteria:

* Any woman with a known allergy to misoprostol or other prostaglandins will be excluded as will any woman under 18 years old (unless she is an emancipated minor)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin | Measured during third trimester and 3-5 days postpartum
  Peri-partum fall in hemoglobin value of over 20% (the outcome of a fall of 2g/dl will also be tested in the pilot) following use of self-administered misoprostol after home birth

SECONDARY OUTCOMES:
Safety | Assessed 3-5 days postpartum
  To assess the safety of ante-natal distribution of misoprostol and its use by women at the time of their home birth, data will be collected on the number of women who report experiencing side effects (including shivering and fever), number of women who are transferred to higher level care, number of women who undergo surgical interventions, number of women who are given blood transfusions, number of maternal deaths, and number of neonatal deaths.
  The exact outcomes as well as the power calculations will only be finalized once the pilot study is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Weeks, Principal Investigator — University of Liverpool
Locations (4):
- Uganda (4):
  - Busiu Health Centre, Mbale, Mbale
  - Lwangoli Health Centre, Mbale, Mbale
  - Mbale Regional Referral Hospital, Mbale, Mbale
  - Siira Health Centre, Mbale, Mbale